CLINICAL TRIAL: NCT04232384
Title: A Randomized Study of "Roll-over' Technique With Standard Abdominal Paracentesis to Improve Cytological Yield in Patients Suspected to Have Peritoneal Carcinomatosis
Brief Title: Comparison of "Roll-over' Technique With Standard Abdominal Paracentesis in Suspected Peritoneal Carcinomatosis
Acronym: ROLLON
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment slow due to COVID-19
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Vishal Sharma, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: NK/6111/DM/055
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Ascites; Peritoneal Carcinomatosis; Peritoneum Neoplasm; Tuberculous Peritonitis
MeSH Terms: conditions — Ascites; Peritoneal Neoplasms; Peritonitis, Tuberculous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard paracentesis group (SPG) (Active Comparator): The patients will be asked to lie supine for 10 minutes and no changes in posture will be allowed for this period. Abdominal paracentesis will be done either by blind technique (in case the ascites is clinically detectable) or ultrasonography-guided (in cases the ascites is not clinically detectable).
  Interventions: Procedure: Standard Paracentesis
- Rollover paracentesis group (ROG) (Experimental): Patients with ascites will be rolled over thrice in bed laterally upto 90 degrees on either side (Figure 1) and ascitic fluid sample is drawn within 1 minute of the last rollover. There will be four steps to this i.e roll over to one side at 90 degrees and then 180 degrees to the other side, then back to the first side and then back to the center (to complete three turns). This will be done after the disinfection and cleaning of the anterior abdominal wall have been done and the personnel involved in the procedure are ready for the paracentesis. The ascitic paracentesis will be initiated within one minute of the completion of the turn. One assistant will maintain a stopwatch during this period to ensure compliance with this.
  Interventions: Procedure: Roll Over Paracentesis

INTERVENTIONS:
Procedure: Standard Paracentesis — The patients will be asked to lie supine for 10 minutes and no changes in posture will be allowed for this period. Abdominal paracentesis will be done either by blind technique (in case the ascites is clinically detectable) or ultrasonography guided (in cases the ascites is not clinically detectable).
  Arms: Standard paracentesis group (SPG)
Procedure: Roll Over Paracentesis — Patients with ascites will be rolled over thrice in bed laterally upto 90 degrees on either side (Figure 1) and ascitic fluid sample is drawn within 1 minute of the last rollover. There will be four steps to this i.e roll over to one side at 90 degrees and then 180 degrees to the other side, then back to the first side and then back to the center (to complete three turns). This will be done after the disinfection and cleaning of the anterior abdominal wall have been done and the personnel involved in the procedure are ready for the paracentesis. The ascitic paracentesis will be initiated within one minute of the completion of the turn. One assistant will maintain a stopwatch during this period to ensure compliance with this.
  Arms: Rollover paracentesis group (ROG)

SUMMARY:
The study will be a randomized trial that will compare two techniques of abdominal paracentesis in patients with suspected peritoneal carcinomatosis. The patients will undergo abdominal paracentesis by the standard technique and a rollover technique. In the standard technique, the patients will lie flat for 10 minutes and abdominal paracentesis will be taken for ascitic fluid cytology. In the rollover group, patients with suspected peritoneal carcinomatosis will be rolled over thrice laterally on each side by 90 degrees and sample will then be obtained for ascitic fluid cytology. both the samples will be processed by blinded cytopathologist for tumour cellularity and diagnostic yield.

DETAILED DESCRIPTION:
Trial Design

The study will be a randomized comparison between two methods of abdominal paracentesis with a cross-over design and each participant will also serve as a control (standard paracentesis).

Participants

The study will be done on the patients who will visit Outpatient departments or admitted as an inpatient in the Post Graduate Institute of Medical Education and Research, Chandigarh.

Screening population: All patients with ascites

Assessment of study population:

Patients fulfilling inclusion and exclusion criteria as per screening will be subjected to baseline investigation in the form of hemogram, biochemistries, coagulogram, ascitic fluid evaluation as per predesigned proforma. All patients in the study group will be subjected to imaging and an attempt will be made to establish the primary site of malignancy based on histopathology.

Patients fulfilling inclusion and exclusion criteria will undergo randomization into two groups. One group will be the standard paracentesis group (SPG) and the other will be the rollover group (ROG). Randomization will be done using an opaque sealed envelope.

Patients fulfilling inclusion and exclusion criteria will undergo abdominal paracentesis twice in one of the following ways.

Standard paracentesis group (SPG):

The patients will be asked to lie supine for 10 minutes and no changes in posture will be allowed for this period. Abdominal paracentesis will be done either by blind technique (in case the ascites is clinically detectable) or ultrasonography-guided (in cases the ascites is not clinically detectable).

Rollover group (ROG):

Patients with ascites will be rolled over thrice in bed laterally up to 90 degrees on either side and the ascitic fluid sample is drawn within 1 minute of the last rollover. There will be four steps to this i.e roll over to one side at 90 degrees and then 180 degrees to the other side and so on to complete three complete turns. This will be done after the disinfection and cleaning of the anterior abdominal wall have been done and the personnel involved in the procedure are ready for the paracentesis. The ascitic paracentesis will be initiated within one minute of the completion of the turn. One assistant will maintain a stopwatch during this period to ensure compliance with this.

Details of ascitic paracentesis

The patient will undergo abdominal paracentesis twice in the order as allocated randomly. The patients will be asked to empty his bladder prior to the procedure. The anterior abdominal wall will be cleaned with a Povidone-iodine solution followed by isopropyl alcohol/ chlorhexidine. The site of the paracentesis will be the peritoneal space in the left lower quadrant between the umbilicus and the anterior superior iliac spine or the patient's flank, depending on the location of the fluid as determined by percussion of the fluid wave. Alternatively, in midline 3 to 4 cm below the umbilicus, halfway between the symphysis pubis and the umbilicus. On both occasions, 20 ml of the ascitic sample will be collected in clean dry containers with appropriate labeling of name and hospital registration number. 20 ml of the sample obtained on each of these occasions will be sent for cytological analysis. To ensure that both the groups are treated similarly the paracentesis will be done using a 20 ml syringe using 21 Gauge 1 1/2" hypodermic needle. It will be ensured to avoid old surgical scars since the bowel may be adherent to the abdominal wall. The site of the paracentesis will be closed with tincture benzoin. The ascitic fluid sample for malignant cytology will be transported to the laboratory within one hour of paracentesis.

ELIGIBILITY:
Inclusion Criteria:

Patient with ascites where a diagnosis of peritoneal carcinomatosis is being considered on the basis of one or more of the following

* Clinical Suspicion of peritoneal carcinomatosis on basis of a history of malignancy, painful ascites and/or loss of weight
* Clinical Suspicion of peritoneal carcinomatosis on the basis of presence of ascites with lump or other stigmata of malignancy
* Suspicion of peritoneal carcinomatosis on imaging suggestive of peritoneal carcinomatosis

Exclusion Criteria:

* Age < 12 years
* Refusal to participate or provide consent
* Evidence of chronic liver disease-related ascites (evidence of cirrhosis on ultrasonography or evidence of portal hypertension eg varices on endoscopy)
* Already diagnosed alternate cause of ascites like cirrhosis, pancreatitis, right heart failure -
* Contraindications to paracentesis in the form of disseminated intravascular coagulation or local site infection.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 71 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Yield of malignant cells | One month
  Number of samples reported positive for malignant cells out of the cases of peritoneal carcinomatosis

SECONDARY OUTCOMES:
Cellularity of the smear of the smear | One day
  Comparison of tumour cellularity, mesothelial cells and inflammatory cells between the two samples will be compared with each other to determine which of the smear had a better cellularity

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Sharma, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma V, Jha DK, Rohilla M, Das CK, Singh H, Irrinki S, Arora A, Saha SC, Gupta P, Mandavdhare HS, Dutta U, Sharma A. 'Rollover' abdominal paracentesis versus standard technique: protocol of a crossover randomized comparative trial. Future Oncol. 2021 Sep;17(26):3425-3431. doi: 10.2217/fon-2020-1050. Epub 2021 Jun 22. PMID 34156308
- [Derived] Jha DK, Rohilla M, Das CK, Irrinki S, Singh H, Arora A, Saha SC, Gupta P, Mandavdhare HS, Dutta U, Sharma A, Sharma V. Randomized crossover trial of 'Roll-over' technique of abdominal paracentesis versus standard technique in suspected malignant ascites. Expert Rev Gastroenterol Hepatol. 2023 Mar;17(3):295-300. doi: 10.1080/17474124.2023.2181785. Epub 2023 Feb 21. PMID 36795510